CLINICAL TRIAL: NCT00428532
Title: The Effect of Licorice Root Extract and Pomegranate Juice on Atherosclerotic Parameters in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009-07-EMC
Record Dates: First submitted 2007-01-27; First posted 2007-01-30 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes Mellitus; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis | interventions — Glycyrrhiza glabra extract

INTERVENTIONS:
Drug: Licorice root extract or Pomegranate juice

SUMMARY:
The study will check whether taking 100 mg of licorice root extract or 250 cc of pomegranate juice daily by men with diabetes mellitus who are non-smokers and already treated with statins decreases the risk of developing atherosclerosis. The hypothesis of the study is that natural anti-oxidants (such as licorice root extract and pomegranate juice), by scavenging free radicals, retard and may even reverse atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Diabetes Mellitus

Exclusion Criteria:

* Younger than 18
* Smoker
* Receiving Fibrates

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-03; Study Completion 2007-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wasseem Rock, MD, Principal Investigator — Ha'Emek Medical Center
Locations (1):
- HaEmek MC, Afula, Israel